CLINICAL TRIAL: NCT06051773
Title: Evaluation of Muscle Involvement in Systemic Sclerosis
Acronym: MUSSc
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Paul DECKER, MD, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI160
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SSc patients
  Interventions: Other: muscle involvement

INTERVENTIONS:
Other: muscle involvement — evaluation of muscle involvement

SUMMARY:
Muscle involvement is poorly described in patients with systemic sclerosis (SSc) .

The prevalence of muscle damage is evaluated at 5-95 % of SSc patients, particularly due to variable definitions depending on the series in the scientific litterature. Muscle clinicobiological and histological presentation an response to immunosuppressive treatments are highly variable. Muscle involvement defined by creatinine kinase (CK) elevation, the presence of electromyography (EMG) abnormalities and/or muscle magnetic resonance imaging (MRI) hyperintensities and/or muscle biopsy inflammation appears to be associated with diffuse SSc, the presence of cardiac damage, and anti-PM-Scl antibodies.

The main objective is to describe muscular manifestations associated with SSc.

Secondary objectives are:

* to compare characteristics between SSc patients with and without muscle involvement
* to determine homogeneous groups of SSc patients with muscle involvement

ELIGIBILITY:
Inclusion Criteria:

* Patients with systemic sclerosis according to 2013 ACR/EULAR classification criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic sclerosis
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with muscle involvement | baseline (J0)
  Muscle involvement is defined by persistent CK elevation, and/or muscle MRI hyperintensities, and/or myogenic abnormalities on EMG, and/or presence of inflammatory myopathy on muscle biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Paul Decker, Nancy, France

IPD SHARING:
Plan to Share IPD: No